CLINICAL TRIAL: NCT00641758
Title: A Double-blind, Randomized, Placebo-controlled, Cross - Over Design, Single Center Study to Evaluate the Effects of Treatment With Pycnogenol® on Endothelial Function in Subjects With Stable Coronary Artery Disease (Pycno2007-003)
Brief Title: Pycnogenol and Endothelial Function in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Prof. Dr. med. Georg Noll, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pycno2007-003
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; endothelial dysfunction; Nitric oxide
MeSH Terms: conditions — Coronary Artery Disease | interventions — pycnogenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pycnogenol (Active Comparator)
  Interventions: Drug: Pycnogenol

INTERVENTIONS:
Drug: Pycnogenol — Pycnogenol 100mg twice daily
  Arms: Pycnogenol
Drug: Placebo — Placebo 100mg twice daily
  Arms: Placebo

SUMMARY:
Pycnogenol® is a proprietary bark extract of the French maritime pine tree (Pinus pinaster ssp. atlantica). Pycnogenol® has prevented pathologic symptoms such as chronic inflammation and increased platelet aggregation, a risk factor for cardiovascular diseases. The endothelium is increasingly recognized not only a target (with vascular remodelling occurring in response to an injury and resulting in atherosclerosis), but also a mediator in the pathogenesis of atherosclerosis. Indeed, endothelial cells play an important regulatory role in the cardiovascular system by the expression of numerous molecules and release of mediators such as nitric oxide (NO), superoxide and endothelin-1 (ET-1). Data from animal studies, as well as human studies indicate that Pycnogenol may improve endothelial function, which is a powerful surrogate for clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease (documented by coronary angiogram, nuclear imaging, positive stress test)
* Stable cardiovascular medication for at least 1 month
* Age ≥ 18 years of age at time of signing the informed consent
* Informed consent for participation in the study

Exclusion Criteria:

* Myocardial infarction, unstable angina, stroke (within 3 months before randomization)
* Thoracic or cardiac surgery and/or coronary intervention/revascularisation procedure (within 3 months before randomization)
* Uncontrolled symptomatic congestive heart failure (NHYA> II) in the last 4 weeks prior to study
* Renal insufficiency (Creatinine Clearance < 50ml/min)
* Ventricular tachyarrhythmias
* Poorly controlled hypertension, defined as resting blood pressure ≥ 160/100 mmHg
* Symptomatic hypotension
* Obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, untreated hypothyroidism or hyperthyroidism and adrenal insufficiency
* Severe uncorrected valvular disease or left ventricular outflow obstruction, which, in the opinion of the investigator, requires surgery
* Long acting nitrates
* Oral or intravenous steroids therapy
* Insulin - dependent diabetes mellitus
* Recipient of any major organ transplant (eg, lung, liver, heart) or renal replacement therapy
* Malignancy (unless healed or remission > 5 years)
* Anaemia (Hb< 10g/dl)
* Known to be human immunodeficiency virus (HIV) positive or active virus - hepatitis
* Alanine transaminase (ALT) or aspartate transaminase (AST) > 3 times the upper limit of the normal range
* Known hypersensitivity to Pycnogenol®
* Alcohol, nicotine abuse or illicit drug abuse
* Pregnancy or breast-feeding, women with child - bearing potential without adequate contraception
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Participation in another study within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the effects of treatment with Pycnogenol® on endothelial function in subjects with stable coronary artery disease. | 8 weeks

SECONDARY OUTCOMES:
Secondary objectives are to evaluate the effect of 8 weeks treatment with Pycnogenol® on inflammation markers, oxidative stress parameters, endothelial progenitor cells, platelet function, 24 hours blood pressure and baroreflex function. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georg Noll, MD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Enseleit F, Sudano I, Periat D, Winnik S, Wolfrum M, Flammer AJ, Frohlich GM, Kaiser P, Hirt A, Haile SR, Krasniqi N, Matter CM, Uhlenhut K, Hogger P, Neidhart M, Luscher TF, Ruschitzka F, Noll G. Effects of Pycnogenol on endothelial function in patients with stable coronary artery disease: a double-blind, randomized, placebo-controlled, cross-over study. Eur Heart J. 2012 Jul;33(13):1589-97. doi: 10.1093/eurheartj/ehr482. Epub 2012 Jan 11. PMID 22240497